CLINICAL TRIAL: NCT02183506
Title: Bioavailability of Both BI 1356 BS and Metformin After Co-administration Compared to the Bioavailability of Multiple Oral Doses of BI 1356 BS 10 mg Daily Alone and Metformin 850 mg Three Times a Day Alone in Healthy Male Volunteers (an Open-label, Randomized, Crossover Study)
Brief Title: Bioavailability of BI 1356 BS and Metformin After Co-administration Compared to the Bioavailability of BI 1356 BS Alone and Metformin Alone in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1218.4
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Metformin; Linagliptin

ARMS (2):
- Metformin (Active Comparator)
  Interventions: Drug: Metformin
- BI 1356 BS and metformin (Experimental): Daily administration of BI 1356 BS alone (day 1 to day 6) followed by the combined treatment of BI 1356 BS with metformin (day 7 to day 9)
  Interventions: Drug: Metformin; Drug: BI 1356 BS

INTERVENTIONS:
Drug: Metformin
Drug: BI 1356 BS
  Arms: BI 1356 BS and metformin

SUMMARY:
Investigate the bioavailability of BI 1356 BS and of metformin after concomitant multiple oral administration of 10 mg BI 1356 BS tablets and 3 x 850 mg metformin in comparison to BI 1356 BS and metformin given alone

ELIGIBILITY:
Inclusion Criteria:

* Healthy males according to the following criteria, based upon a complete medical history, including the physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), clinical laboratory tests

  * No finding deviating from normal and of clinical relevance
  * No evidence of a clinically relevant concomitant disease
* Age ≥ 21 and Age ≤ 50 years
* BMI (Body Mass Index) ≥ 18.5 and ≤ 29.9 kg/m2
* Ability to give signed and dated written informed consent prior to admission to the study in accordance with good clinical practice (GCP) and the local legislation

Exclusion Criteria:

* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial by the investigator
* Intake of drugs with a long half-life (>24 hours) within one month or less than 10 half-lives of the respective drug prior to administration or during the conduct of this trial (review with clinical monitor if there is a question)
* Use of drugs which might reasonably influence the results of the trial (based on knowledge at the time of protocol preparation) within 10 days prior to administration or during the conduct of this trial
* Participation in another trial with an investigational drug within two months prior to administration or during the conduct of this trial
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking during the conduct of this trial
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the conduct of this trial)
* Excessive physical activities (within one week prior to administration or during the conduct of this trial)
* Any laboratory value outside the normal reference range that is of clinical relevance
* Inability to comply with the dietary regimen of the study center
* No adequate contraception (condom use plus another form of contraception e.g., spermicide, oral contraceptive taken by female partner, sterilization) during the whole study period from the time of the first intake of study drug until one month after the last intake of drug

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2005-09; Primary Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve (AUC) of the analytes in plasma at different time points | up to 240 hours after start of treatment
Maximum concentration (Cmax) of the analytes in plasma at different time points | up to 240 hours after start of treatment

SECONDARY OUTCOMES:
Time from last dosing to maximum concentration of the analytes in plasma at steady state (tmax,ss) | up to 240 hours after start of treatment
Minimum concentration of the analytes in plasma at steady state (Cmin,ss) over a uniform dosing interval τ | up to 240 hours after start of treatment
Terminal rate constant of the analytes in plasma at steady state (λz,ss ) | up to 240 hours after start of treatment
Terminal half-life of the analytes in plasma at steady state (t1/2,ss ) | up to 240 hours after start of treatment
Mean residence time of the analytes in the body at steady state after oral administration (MRTpo,ss) | up to 240 hours after start of treatment
Apparent clearance of the analytes in the plasma at steady state (CL/F,ss) following extravascular multiple dose administration | up to 240 hours after start of treatment
Apparent volume of distribution during the terminal phase λz at steady state (Vz/F,ss) following extravascular administration | up to 240 hours after start of treatment
Measurements of dipeptidylpeptidase 4 (DPP-IV) activity | up to 240 hours after start of treatment
Number of patients with adverse events | up to 60 days
Number of patients with clinically abnormal changes in laboratory values | Baseline, up to 14 days after last drug administration
Number of patients with clinically relevant changes in vital signs | Baseline, up to 14 days after last drug administration
feτ,ss (fraction of the dose excreted unchanged in urine at steady state) | 0-4 h, 4-8 h, 8-12 h and 12-24 hours after drug administration on days 3, 6, 9
CLR,ss (renal clearance of the analyte in plasma at steady state) | 0-4 h, 4-8 h, 8-12 h and 12-24 hours after drug administration on days 3, 6, 9